CLINICAL TRIAL: NCT05667233
Title: A Pilot Study Examining Differences in Waist, Upper-arm, Mid-thigh Circumference and Body Composition When Training to Momentary Muscular Fatigue Versus Close Failure-proximity Amongst Healthy Male Biological Sex University-aged Students
Brief Title: Examining Changes in Muscle Size and Body Composition Between Two Hypertrophy Resistance Training Programs in Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, Jeffery Zahavich, PhD, Instructor, Kinesiology, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-6399
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Hypertrophy; Body Weight Changes; Muscle Size
Keywords: Exercise; Resistance Training
MeSH Terms: conditions — Hypertrophy; Body Weight Changes; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups (train to failure OR train to non-failure) and stratified according to their recent training experience (beginner [3-9 months experience], intermediate [9-18 months experience], advanced [>18 months experience]).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Train to failure (Active Comparator): Training regime will be highly uncomfortable since it will be both physically and psychologically challenging to push to momentary muscular fatigue (MMF; i.e., failure).
  Interventions: Other: Resistance Training Program
- Train to non-failure (Active Comparator): Training regime will be moderately uncomfortable as participants will be training at a close proximity to failure (4-0 repetitions in reserve; i.e., non-failure).
  Interventions: Other: Resistance Training Program

INTERVENTIONS:
Other: Resistance Training Program — Participants will undergo a high exertion machine-based resistance training protocol.

SUMMARY:
This study aims to investigate if a less physically and psychologically taxing approach to resistance training can generate equal or greater outcomes when compared to a more physically and psychologically taxing approach.

DETAILED DESCRIPTION:
Resistance training is commonly used to improve body composition, gain strength, increase muscle size (i.e., hypertrophy) and prevent muscle atrophy (i.e., muscle wasting). The most optimal mode of building muscle remains unclear, however there are many mechanisms that can be tested to yield optimal results. One variable that can be manipulated when designing a hypertrophy-focused resistance training regimen is intensity (i.e., proximity-to-failure). Proximity-to-failure is defined as the number of repetitions remaining in a set of prescribed exercises prior to reaching momentary muscular failure (MMF). MMF is when an individual cannot complete the lowering or concentric phase of a given repetition with a full range-of-motion without deviation from the prescribed form of the exercise. For all lifters, particularly amongst older populations, it can be psychologically demanding to push to MMF, and may increase the risk of delayed onset muscle soreness (DOMS) and/or injury due to technical breakdown. In contrast, there is some evidence that suggests training to a slightly less intensity (i.e., within 1-4 repetitions in reserve [RIR]) may result in comparable hypertrophic results with less of a physical and psychological demand on participants.

For these reasons, this study looks to investigate if an easier (i.e., less intense) approach to training such as training with repetitions in reserve (RIR), warrants similar or better muscle hypertrophy adaptations to MMF.

ELIGIBILITY:
Inclusion Criteria:

* biological male
* age 18 years or older
* enrolled at Dalhousie university
* minimum 3-months of consistent (at least 2x/week) resistance training experience

Exclusion Criteria:

* body fat percentage 25% or greater (obese)
* use of performance enhancing drugs that aim to increase rate of muscle growth (i.e., androgenic steroids, anabolic steroids, selective androgen receptive modulators, growth hormone).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Segment girth (cm) | 8-weeks
  Upper arm (biceps) circumference, mid-thigh (quadriceps) circumference, waist (abdomen) circumference

SECONDARY OUTCOMES:
Body composition (kg) | 8-weeks
  Fat mass, Fat-free mass, Total Body Mass (fat mass + fat free mass)
Body Fat Percentage | 8-weeks
  Fat Mass (kg) / Total Body mass (kg) * 100

CONTACTS AND LOCATIONS:
Locations (1):
- Dalplex Fitness Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No